CLINICAL TRIAL: NCT05038709
Title: Does the Addition of a Traction Pad Reduce the Rate of Postoperative Pudendal Neuralgia?
Brief Title: Positioning for Hip Arthroscopic Surgery to Reduce Postoperative Numbness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Vehniah Tjong, Assistant Professor of Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00214620
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Hip Osteoarthritis; Hip Injuries; Hip Sprain; Hip Strain
Keywords: arthroscopy; traction
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pink Pad (Experimental): Hip arthroscopy using The Pink Pad Hip Kit Patient Positioning System (Xodus Medical, New Kensington, PA). The pad is placed between the patient and the traction table, using a perineal post.
  Interventions: Device: The Pink Pad Hip Kit
- Control (No pad) (No Intervention): Hip arthroscopy in the usual fashion, no pad, using traction table with perineal post.

INTERVENTIONS:
Device: The Pink Pad Hip Kit — The pad is placed between the patient and the traction table to reduce pressure to the pudendal nerve exerted by the perineal post.
  Other Names: Xodus Medical
  Arms: Pink Pad

SUMMARY:
Compared to the knee and shoulder, the hip joint leaves relatively little space to maneuver arthroscopic instruments and camera. To expand the potential space in the hip joint, traction is commonly applied to the operative leg through a perineal post. This is an effective technique to improve the working space for arthroscopy, however it has been associated with complications, including perineal numbness. Traction pads, used alone or with a perineal post, can reduce pressure on the perineal area, thus reducing numbness. The investigators hypothesize that positioning hip arthroscopy patients using a traction pad on a standard traction table with a perineal post will reduce the incidence and duration of postoperative perineal numbness.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Northwestern Memorial Hospital (NMH) or to a Northwestern orthopaedic surgery faculty member's clinic undergoing hip arthroscopy
* Ability to read and speak English

Exclusion Criteria:

* Revision surgery
* Oncologic surgery
* Use of regional anesthesia
* Arthroscopic hip surgery that involves procedures other than labral repair, acetabuloplasty, CAM-plasty, IT band windowing, Iliopsoas lengthening

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
patient-reported post-operative numbness | Baseline prior to surgery
  Y/N Are you experiencing complete or partial numbness prior to your surgery?
patient-reported post-operative numbness | 72 hours after surgery
  Y/N Are you experiencing complete or partial numbness as a result of your surgery?
patient-reported numbness | 1 week after surgery
  Y/N Are you experiencing complete or partial numbness as a result of your surgery?
patient-reported numbness | 3 weeks after surgery
  Y/N Are you experiencing complete or partial numbness as a result of your surgery?
patient-reported numbness | 6 weeks after surgery
  Y/N Are you experiencing complete or partial numbness as a result of your surgery?

SECONDARY OUTCOMES:
patient-reported difficulty urinating | Baseline prior to surgery
  Y/N Have you experienced difficulty urinating?
patient-reported difficulty urinating | 72 hours after surgery
  Y/N Have you experienced difficulty urinating?
patient-reported difficulty urinating | 1 week after surgery
  Y/N Have you experienced difficulty urinating?
patient-reported difficulty urinating | 3 weeks after surgery
  Y/N Have you experienced difficulty urinating?
patient-reported difficulty urinating | 6 weeks after surgery
  Y/N Have you experienced difficulty urinating?
patient-reported difficulty with bowel movements | Baseline prior to surgery
  Y/N Have you experienced difficulty with bowel movements?
patient-reported difficulty with bowel movements | 72 hours after surgery
  Y/N Have you experienced difficulty with bowel movements?
patient-reported difficulty with bowel movements | 1 week after surgery
  Y/N Have you experienced difficulty with bowel movements?
patient-reported difficulty with bowel movements | 3 weeks after surgery
  Y/N Have you experienced difficulty with bowel movements?
patient-reported difficulty with bowel movements | 6 weeks after surgery
  Y/N Have you experienced difficulty with bowel movements?
patient-reported skin changes or breakdown | Baseline prior to surgery
  Y/N Have you experienced skin changes or skin breakdown?
patient-reported skin changes or breakdown | 72 hours after surgery
  Y/N Have you experienced skin changes or skin breakdown?
patient-reported skin changes or breakdown | 1 week after surgery
  Y/N Have you experienced skin changes or skin breakdown?
patient-reported skin changes or breakdown | 3 weeks after surgery
  Y/N Have you experienced skin changes or skin breakdown?
patient-reported skin changes or breakdown | 6 weeks after surgery
  Y/N Have you experienced skin changes or skin breakdown?
patient-reported sexual disfunction or erectile disfunction | Baseline prior to surgery
  Y/N Have you experienced sexual dysfunction/erectile dysfunction?
patient-reported sexual disfunction or erectile disfunction | 72 hours after surgery
  Y/N Have you experienced sexual dysfunction/erectile dysfunction?
patient-reported sexual disfunction or erectile disfunction | 1 week after surgery
  Y/N Have you experienced sexual dysfunction/erectile dysfunction?
patient-reported sexual disfunction or erectile disfunction | 3 weeks after surgery
  Y/N Have you experienced sexual dysfunction/erectile dysfunction?
patient-reported sexual disfunction or erectile disfunction | 6 weeks after surgery
  Y/N Have you experienced sexual dysfunction/erectile dysfunction?

CONTACTS AND LOCATIONS:
Overall Officials: Vehniah K Tjong, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Orthopaedic Surgery, Chicago, Illinois, United States